CLINICAL TRIAL: NCT00214214
Title: A Pilot Study to Determine the Safety of Campath-1H (Anti-CD52 Antibody) Therapy in Newly Diagnosed Subjects With Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-2003-0405
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: New Onset Type 1 Diabetes Mellitus
MeSH Terms: interventions — Alemtuzumab

INTERVENTIONS:
Drug: Campath 1H® (Alemtuzumab)

SUMMARY:
The rationale for the study is to determine if Campath-1H can be used in patients recently diagnosed with type I DM, to induce a state of immunological unresponsiveness such that subjects can safely preserve beta cell mass and eliminate or lower insulin requirements, preserving excellent metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ages 18-35, with new onset type 1 diabetes mellitus (within 2-12 weeks of diagnosis), one or more islet autoantibody to GAD, IA2, IAA or islet cell cytoplasmic antibody (ICA) within 2 weeks of diabetes diagnosis.

Exclusion Criteria:

* Subjects under 18 years of age or over 35 years of age.
* Subjects who have previously received an organ transplant.
* Subjects who are currently receiving systemic corticosteroids for other medical diseases in which the physician feels discontinuation of corticosteroids is contraindicated.
* Subjects with a history of other medical condition(s) known to affect blood glucose values (i.e., Cushing's disease, acromegaly).
* Subjects with a history of other chronic systemic inflammatory or autoimmune disease or other severe medical condition. (A history of treated hypothyroidism with documentation of normal serum thyroid hormone levels will not be exclusionary.)
* Patients with a history of hepatitis B, hepatitis C, or HIV.
* PPD positive at the time of evaluation.
* Thrombocytopenia or neutropenia. Individuals will be considered to have thrombocytopenia if they have a platelet count <100,000 platelets/mm2 or <3,000 WBC/ml.
* Subjects with a history of renal, pulmonary, or cardiac failure
* Subjects with severe systemic infections. Only those subjects who have completed treatment and have shown a complete clinical resolution will be considered eligible for the study.

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10

PRIMARY OUTCOMES:
to determine if Campath-1H can be used in patients recently diagnosed with type I DM

SECONDARY OUTCOMES:
to determine if Campath-1H can eliminate or lower insulin requirements

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernandez, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States